CLINICAL TRIAL: NCT04285047
Title: Advancing the Patient Experience in Chronic Obstructive Pulmonary Disease (APEX COPD)
Acronym: APEX COPD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Optimum Patient Care (Other)
Collaborators: Boehringer Ingelheim (Industry); DARTNet Institute (Other Government); American Academy of Family Physicians National Research Network (AAFP NRN) (Unknown); Respiratory Effectiveness Group (Other)
Responsible Party: Sponsor
Other Study IDs: OPCG -1803
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (13645005)
Keywords: Chronic Obstructive Pulmonary Disease; Chronic Obstructive Lung Disease; Chronic Obstructive Airway Disease; Registry; Electronic Health Record; Electronic Medical Record; Patient Reported Information and Outcomes; Treatment; Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Advancing Patient Experience (APEX) in COPD — Involves both EMR and PRIO data

SUMMARY:
APEX COPD is registry to provide a mechanism to standardize, store and utilize data to enable greater power to answer key research questions, and to improve patient outcomes in COPD primary care.

DETAILED DESCRIPTION:
In the process of creating of a high-quality longitudinal dataset combining COPD templates and patient reported information and outcome (PRIO) to evaluate outcomes the APEX COPD registry supports changes and improvements in medical practice and deliver high quality research through the following mechanisms:

* Templates integrated into the primary care clinical systems to support standardization of care and data over time.
* Informing doctors at the point of consultation about the status of their patients through data-driven feedback.
* Pre-filled electronic data templates from existing EHR data and questionnaires to reduce administrative burden for Primary Care Clinicians (PCC).
* Engaging primary care clinicians in ongoing quality improvement initiatives directly at the point of care.
* Research publications regarding treatment effectiveness and associated risk in mild to moderate COPD, reason for therapy switch/escalation and hidden undiagnosed and untreated COPD patients in primary care.
* A strong network of primary care clinicians caring for patients with COPD in the US to drive the initiative and ensure impact on clinical practice through educational events, academic organizations and research outputs.

The APEX COPD steering committee (SC) comprise of collective clinical expertise, scientific knowledge and experience in EHR, databases and research, forming an essential element of the APEX COPD registry. The SC plays an essential role in the development and governance of the APEX COPD registry, representing the sites participating, and providing the expertise necessary to implement and drive the initiative. Within this committee a smaller management group guides the operational aspects of the registry.

The research database uses the Observational Medical Outcomes Partnership (OMOP) v5 Common Data Model (CDM) and the OMOP terminology will be updated at least bi-annually. Standardized OMOP Concept IDs will utilize SNOMED, RxNorm and may be adjusted to improve data compatibility with other OPC COPD databases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic code for COPD or COPD monitoring review code prior to or at consultation
* Aged ≥35 years at COPD diagnosis

Exclusion Criteria:

* Patients receiving hospice care
* Patients being actively treated for a cancer diagnosis (not skin)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study populations comprise of patients aged over 35 years and receiving care for COPD at participating primary care sites across the US in accordance with local regulatory/ethical requirements.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2019-03-23 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Describe and characterize the COPD primary care patient population's natural history | 31 December 2018 to 31 December 2022
  Baseline data from electronic health record (EHR) and patient reported information and outcomes (PRIO). The EHR data will be updated every three months.
Evaluate the comparative clinical, safety and cost effectiveness of current COPD treatments by class of therapy for COPD overall and in specific patient groups/phenotypes, to understand the predictors of response to available COPD treatment options | 31 December 2018 to 31 December 2022
  Patient reported information and outcomes (PRIO) will be collected annually and before very visit to their doctor

SECONDARY OUTCOMES:
Improve quality of care, and primary care patient outcomes | 31 December 2018 to 31 December 2022
Understand the clinical phenotypes | 31 December 2018 to 31 December 2022
Understand the current burden and minimize side effects | 31 December 2018 to 31 December 2022
Support the development of effective and efficient diagnostic routines | 31 December 2018 to 31 December 2022
comparing clinician-diagnosed COPD at baseline against established | 31 December 2018 to 31 December 2022
Describe disease management pattern | 31 December 2018 to 31 December 2022
Assess impact of inhaler technique | 31 December 2018 to 31 December 2022
Describe factors associated with treatment choice at baseline | 31 December 2018 to 31 December 2022
Describe risk factors | 31 December 2018 to 31 December 2022
Assess the occurrence of exacerbations and other conditions | 31 December 2018 to 31 December 2022
Assess biomarker data and estimate their predictive value for disease diagnosis | 31 December 2018 to 31 December 2022
identify patients who may be eligible for participation in future research studies | 31 December 2018 to 31 December 2022

CONTACTS AND LOCATIONS:
Overall Officials: Wilson D Pace, MD, Principal Investigator — Professor
Locations (4):
- United States (4):
  - Miramont Family Medicine, Fort Collins, Colorado
  - Urban Family Practice, Buffalo, New York
  - MetroHealth System, Cleveland, Ohio
  - Bandera Family Health Care, San Antonio, Texas